CLINICAL TRIAL: NCT07334470
Title: The BRAVE Study: A Sensitivity Intervention With Nursing Students Using Simulation
Brief Title: Weight Bias Reducation Intervention With Nursing Students Using Simulation: The BRAVE Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Villanova University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2025-30
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Weight Bias
Keywords: weight bias; nursing education; obesity
MeSH Terms: conditions — Weight Prejudice; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRAVE Intervention (Experimental): BRAVE (Building Respect and Acceptance through Valuing Everybody). Participants will receive two 30-minute Simulated Patients (SP) encounters: 1 at baseline (before the weight bias or obesity presentations) and one at 1.5 months after the initial education. The simulation encounters will include SPs living with higher body weight and will emphasize communication skills to prevent weight bias in the clinical environment. BRAVE arm will consist of two educational sessions focused on reducing weight bias in health care. Both BRAVE SP encounters will provide a Debriefing for Meaningful Learning segment tailored to focus on reducing weight bias.
  Interventions: Behavioral: BRAVE
- SOL (Placebo Comparator): SOL (Standard Obesity Lecture). The control arm will experience two standard obesity lectures and two simulation encounters with standardized patients living with higher body weight. The control condition consists of two sessions, each of which includes a one-hour presentation on obesity. Both simulations will be followed by standard Debriefing for Meaningful Learning segments, but these segments will focus only on the medical conditions and risk factors of obesity and no feedback on communication skills will be provided.
  Interventions: Behavioral: SOL: Standard Obesity Lecture

INTERVENTIONS:
Behavioral: BRAVE — In addition to the two simulation encounters, the BRAVE arm will include an initial one-hour educational presentation on weight bias in health care; prevalence, and influences of weight bias on health/health care, factors affecting obesity, approaching weight-related discussions with patients with sensitivity and empathy, and effective communication strategies. Clinical communication behaviors will also be taught, such as asking permission, using non-stigmatizing language, and engaging in judgment-free weight-related discussions with patients. They will also have role-play and case-study scenarios to integrate and practice the communication strategies. Following the second simulation and DML, students in the BRAVE arm will participate in a continuation of the weight bias reduction education including concepts of Motivational Interviewing, Shared Decision Making, and weight management conversations to prevent weight bias in the clinical environment.
  Arms: BRAVE Intervention
Behavioral: SOL: Standard Obesity Lecture — SOL: (Standard Obesity Lecture) SOL arm education will include a presentation on obesity as a disease, its prevalence, causes, health risks, psychological and socioeconomic impact, and a standard obesity assessment. Following the second simulation, students in the SOL groups will participate in a continuation of the standard obesity education to build on concepts from session 1. The second presentation will be a recap on weight management in clinical practice. Readings will focus on the medical consequences of obesity, and the economic cost of obesity. Both Debriefing for Meaningful Learning segments will focus on the disease itself and not include components of obesity or body weight.
  Arms: SOL

SUMMARY:
This randomized controlled trial will be a curriculum-embedded weight sensitivity training program. There will be two groups. The control group will receive the standard obesity lecture (SOL) and the intervention group will receive the BRAVE Intervention (BRAVE: Building Respect and Acceptance through Valuing Everybody); a Weight Bias Reduction (WBR) intervention. Both groups will have two simulation encounters with standardized patients who are living with obesity and the outcome will be to improve weight bias and increase weight sensitivity over one year. Participants will include second- and fourth-year nursing students. Two cohorts of nursing students will be recruited over two years during orientation for their NUR courses (n = 368); a combined total of 420 students are typically enrolled in these courses. Study participants will be randomized by 8-person simulation groups (clusters) to either the BRAVE intervention or SOL control group. They will then participate in the two simulation-based experiences and weight bias reduction education or standard obesity lecture, respectively, with a debriefing segment and educational components. To compare the efficacy of BRAVE groups to SOL groups in validated questionnaires will assess changing attitudes, beliefs, and clinical communication behaviors when comparing baseline to 3 months post-intervention, and one year after the intervention.

DETAILED DESCRIPTION:
Longstanding evidence documents the detrimental effects of provider biases on poor patient outcomes. Weight bias among nurses is an understudied concept that causes increased morbidity and mortality in populations living with obesity. Specifically, studies show that nurses with weight bias: 1) assume patients' symptoms are related to obesity and do not further probe underlying causes, 2) are more reluctant to perform preventative health screenings (such as pelvic examinations, cancer screenings, and mammograms), 3) spend less time engaging with patients during visits, all of which causes patients to withdraw from the provider, potentially resulting in difficulty remembering or adhering to provider advice and avoiding future preventative care visits.

Given the increasing rates of obesity in the United States, efforts are direly needed to improve the care provided by nurses who work with this demographic to thwart preventable health consequences (e.g., diabetes, heart disease). Our previous research showed favorable improvements in nursing students' attitudes and beliefs toward individuals with obesity following a Weight Bias Reduction (WBR) intervention when implemented into their clinical course. Gaps remain, however, in 1) whether WBR interventions can translate into behavior change in clinical practice and make notable reductions in the weight bias patients are experiencing, and 2) whether these changes are sustained over time. To fill these gaps, the proposed BRAVE (Building Respect and Acceptance through Valuing Everybody, WBR intervention) will build on our previous research to include education on communication skills and empathic competence, as well as utilize simulation with standardized participants living with obesity.

The study design is a cluster-randomized controlled trial comparing BRAVE to SOL (Standard Obesity Lecture) in reducing weight bias among nursing students (n = 368) and will include follow-up measures to determine the intervention's sustained effects one year later. Additionally, the broader impacts of this BRAVE intervention can enhance long-term health outcomes with the potential for improved patient satisfaction while navigating the healthcare system.

AIM 1: To compare the efficacy of BRAVE groups to SOL groups in changing attitudes, beliefs, and clinical communication behaviors when comparing baseline to 3 months post-intervention.

Hypothesis 1: BRAVE groups will demonstrate statistically significant improvements in attitudes, beliefs, and clinical communication behaviors that are greater than those of SOL groups when comparing baseline and 3 months post-intervention.

* Attitudes will be measured by Attitudes Towards Higher Weight Persons (ATOP-HW) Questionnaire scores.
* Beliefs will be measured by Beliefs About Obese Persons (BAOP) Questionnaire scores.
* Clinical Communication Behaviors will be measured by SE-12, WSI, and SEGUE scores.

AIM 2: To evaluate whether changes in attitudes, beliefs, and clinical communication behaviors between BRAVE and SOL groups are sustained over a one-year period.

Hypothesis 2: BRAVE groups will sustain statistically significant improvements in attitudes, beliefs, and clinical communication behaviors toward obesity compared to SOL groups when assessed from Session 2 to Session 3 one year post-intervention.

Attitudes will be measured by Attitudes Towards Higher Weight Persons (ATOP-HW) Questionnaire scores.

Beliefs will be measured by the Beliefs About Obese Persons (BAOP) Questionnaire scores.

Clinical Communication Behaviors (self-efficacy) will be measured by the SE-12 scores.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students aged 18-25
* Nursing students during their second or fourth year of the traditional or FLEX BSN undergraduate curriculum (in specified nursing courses)

Exclusion Criteria:

* Non-nursing students
* Nursing students taking courses out of the normal curriculum sequence
* Nursing students who are not of traditional undergraduate ages (18-25 years)
* Students who decline to consent

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 368 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2028-05-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Attitudes Towards Higher Weight Persons (ATOP-HW) | Baseline to 3 Months
  Estimated Mean Change Score.The ATOP-HW is a 20-item Likert rating scale that focuses on perceptions and attitudes about people living with obesity. Higher scores reflect more positive attitudes toward persons with obesity.
Beliefs About Obese Persons Scale (BAOP) | Baseline to 3 Months
  The BAOP is an eight-item Likert rating scale that assesses beliefs about the causes of obesity. Each question asks individuals to indicate the extent of agreement or disagreement (+3 to -3) to a specific statement, such as "obesity is really caused by a lack of willpower." Higher scores indicate beliefs that obesity is not controllable.
SE-12 (Self-Efficacy) Scale | Baseline to 3 Months
  The SE-12 is a 12-item questionnaire assessing self-efficacy by clinicians in clinical communications.

SECONDARY OUTCOMES:
SEGUE Framework | Baseline and 3 Months
  The SEGUE Checklist is a valid and reliable checklist designed to be used in various settings to teach, assess, and improve communication skills with medical providers.The SEGUE acronym stands for Set the Stage, Elicit information, Give information, Understand the patient's perspective, and End the encounter. SEGUE includes a 25-item dichotomous checklist to evaluate whether a task was completed.
Weight Sensitivity Instrument (WSI) | Baseline and 3 Months
  The WSI is a 15-item checklist that will assess aspects of physical assessment skills, patient psychological safety, and weight sensitivity of the session.
Attitudes Towards Higher Weight Persons (ATOP-HW) Questionnaire | Baseline to 1 Year; 3 months to 1 Year
  The ATOP-HW is a 20-item Likert rating scale that focuses on perceptions and attitudes about obese people. Higher scores reflect more positive attitudes toward persons with obesity.
Beliefs About Obese Persons Scale (BAOP) | Baseline to 1 Year; 3 months to 1 year
  The BAOP is an eight-item Likert rating scale that assesses beliefs about the causes of obesity. Each question asks individuals to indicate the extent of agreement or disagreement (+3 to -3) to a specific statement, such as "obesity is really caused by a lack of willpower." Higher scores indicate beliefs that obesity is not controllable
SE-12 (Self-Efficacy) Questionnaire | Baseline to 1 year; 3 months to 1 year
  The SE-12 is a 12-item questionnaire assessing self-efficacy by clinicians in clinical communications.

CONTACTS AND LOCATIONS:
Locations (1):
- Villanova University, Villanova, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geller G, Watkins PA. Addressing Medical Students' Negative Bias Toward Patients With Obesity Through Ethics Education. AMA J Ethics. 2018 Oct 1;20(10):E948-959. doi: 10.1001/amajethics.2018.948. PMID 30346923
- [Background] Gayer GG, Weiss J, Clearfield M. Fundamentals for an Osteopathic Obesity Designed Study: The Effects of Education on Osteopathic Medical Students' Attitudes Regarding Obesity. J Am Osteopath Assoc. 2017 Aug 1;117(8):495-502. doi: 10.7556/jaoa.2017.099. PMID 28759091
- [Background] Charlesworth TES, Banaji MR. Patterns of Implicit and Explicit Attitudes: I. Long-Term Change and Stability From 2007 to 2016. Psychol Sci. 2019 Feb;30(2):174-192. doi: 10.1177/0956797618813087. Epub 2019 Jan 3. PMID 30605364
- [Background] Bell ML, Rabe BA. The mixed model for repeated measures for cluster randomized trials: a simulation study investigating bias and type I error with missing continuous data. Trials. 2020 Feb 7;21(1):148. doi: 10.1186/s13063-020-4114-9. PMID 32033617
- [Background] Makoul G. The SEGUE Framework for teaching and assessing communication skills. Patient Educ Couns. 2001 Oct;45(1):23-34. doi: 10.1016/s0738-3991(01)00136-7. PMID 11602365
- [Background] Axboe MK, Christensen KS, Kofoed PE, Ammentorp J. Development and validation of a self-efficacy questionnaire (SE-12) measuring the clinical communication skills of health care professionals. BMC Med Educ. 2016 Oct 18;16(1):272. doi: 10.1186/s12909-016-0798-7. PMID 27756291
- [Background] Allison, D.B., Basile, V.C., & Yuker, H.E. (1991). The measurement of attitudes toward and beliefs about obese persons. International Journal of Eating Disorders, 10(5). 599-607
- [Background] Dreifuerst, K. T. (2015). Getting started with debriefing for meaningful learning. Clinical Simulation in Nursing, 11(5), 268-275. http://dx.doi.org/10.1016/j.ecns.2015.01.005
- [Background] Douglas, V.J., Kwan, M.Y., Minnich, A.M., Converse, J.N., Wonderlich, J.A., & Gordon, K.H. (2022). An examination of the link between empathy and weight-based victimization. Social Sciences & Humanities Open, 5(1), 100247 https://doi.org/10.1016/j.ssaho.2022.100247
- [Background] Burke SE, Dovidio JF, Przedworski JM, Hardeman RR, Perry SP, Phelan SM, Nelson DB, Burgess DJ, Yeazel MW, van Ryn M. Do Contact and Empathy Mitigate Bias Against Gay and Lesbian People Among Heterosexual First-Year Medical Students? A Report From the Medical Student CHANGE Study. Acad Med. 2015 May;90(5):645-51. doi: 10.1097/ACM.0000000000000661. PMID 25674910
- [Background] Dovidio, J.F., Gaertner, S.L., & Kawakami, K. (2003). Intergroup contact: the past, present, and future. Group Process Intergroup Relations, 6, 5-21.
- [Background] Pettigrew TF, Tropp LR. A meta-analytic test of intergroup contact theory. J Pers Soc Psychol. 2006 May;90(5):751-83. doi: 10.1037/0022-3514.90.5.751. PMID 16737372
- [Background] Allport, G.W. (1954). The Nature of Prejudice, Reading, Massachusetts: Addison-Wesley
- [Background] Phelan SM, Puhl RM, Burgess DJ, Natt N, Mundi M, Miller NE, Saha S, Fischer K, van Ryn M. The role of weight bias and role-modeling in medical students' patient-centered communication with higher weight standardized patients. Patient Educ Couns. 2021 Aug;104(8):1962-1969. doi: 10.1016/j.pec.2021.01.003. Epub 2021 Jan 5. PMID 33487507
- [Background] Kushner RF, Zeiss DM, Feinglass JM, Yelen M. An obesity educational intervention for medical students addressing weight bias and communication skills using standardized patients. BMC Med Educ. 2014 Mar 18;14:53. doi: 10.1186/1472-6920-14-53. PMID 24636594
- [Background] Clinton AJ, Pollini RA. Using Positive Empathy Interventions to Reduce Stigma Toward People Who Inject Drugs. Front Psychol. 2021 Jul 9;12:616729. doi: 10.3389/fpsyg.2021.616729. eCollection 2021. PMID 34305698
- [Background] Hunter J, Rawlings-Anderson K, Lindsay T, Bowden T, Aitken LM. RETRACTED: Exploring student nurses' attitudes towards those who are obese and whether these attitudes change following a simulated activity. Nurse Educ Today. 2018 Jun;65:225-231. doi: 10.1016/j.nedt.2018.03.013. Epub 2018 Mar 22. PMID 29604606
- [Background] Barra M, Singh Hernandez SS. Too big to be seen: Weight-based discrimination among nursing students. Nurs Forum. 2018 Oct;53(4):529-534. doi: 10.1111/nuf.12282. Epub 2018 Jul 3. PMID 29968365
- [Background] Moore CH, Oliver TL, Randolph J, Dowdell EB. Interventions for reducing weight bias in healthcare providers: An interprofessional systematic review and meta-analysis. Clin Obes. 2022 Dec;12(6):e12545. doi: 10.1111/cob.12545. Epub 2022 Aug 10. PMID 35946476
- [Background] Danielsdottir S, O'Brien KS, Ciao A. Anti-fat prejudice reduction: a review of published studies. Obes Facts. 2010 Feb;3(1):47-58. doi: 10.1159/000277067. Epub 2010 Feb 11. PMID 20215795
- [Background] Diedrichs PC, Barlow FK. How to lose weight bias fast! Evaluating a brief anti-weight bias intervention. Br J Health Psychol. 2011 Nov;16(4):846-61. doi: 10.1111/j.2044-8287.2011.02022.x. Epub 2011 Apr 8. PMID 21988068
- [Background] Balkhi, A.M., Parent, M.C., & Mayor, M. (2013) Impact of Perceived Weight Discrimination on Patient Satisfaction and Physician Trust, Fat Studies, 2(1), 45-55, DOI: 10.1080/21604851.2013.731955
- [Background] Alberga AS, Edache IY, Forhan M, Russell-Mayhew S. Weight bias and health care utilization: a scoping review. Prim Health Care Res Dev. 2019 Jul 22;20:e116. doi: 10.1017/S1463423619000227. PMID 32800008
- [Background] Rubino F, Puhl RM, Cummings DE, Eckel RH, Ryan DH, Mechanick JI, Nadglowski J, Ramos Salas X, Schauer PR, Twenefour D, Apovian CM, Aronne LJ, Batterham RL, Berthoud HR, Boza C, Busetto L, Dicker D, De Groot M, Eisenberg D, Flint SW, Huang TT, Kaplan LM, Kirwan JP, Korner J, Kyle TK, Laferrere B, le Roux CW, McIver L, Mingrone G, Nece P, Reid TJ, Rogers AM, Rosenbaum M, Seeley RJ, Torres AJ, Dixon JB. Joint international consensus statement for ending stigma of obesity. Nat Med. 2020 Apr;26(4):485-497. doi: 10.1038/s41591-020-0803-x. Epub 2020 Mar 4. PMID 32127716
- [Background] Lumley E, Homer CV, Palfreyman S, Shackley P, Tod AM. A qualitative study to explore the attitude of clinical staff to the challenges of caring for obese patients. J Clin Nurs. 2015 Dec;24(23-24):3594-604. doi: 10.1111/jocn.13016. Epub 2015 Oct 14. PMID 26467348
- [Background] Tanneberger A, Ciupitu-Plath C. Nurses' Weight Bias in Caring for Obese Patients: Do Weight Controllability Beliefs Influence the Provision of Care to Obese Patients? Clin Nurs Res. 2018 May;27(4):414-432. doi: 10.1177/1054773816687443. Epub 2017 Jan 4. PMID 28052689
- [Background] Pervez, H., & Ramonaledi, S. (2017) Nurses' attitudes towards obese patients: a review of the literature. Nursing Times, 113(2), 42-45.
- [Background] Brown I. Nurses' attitudes towards adult patients who are obese: literature review. J Adv Nurs. 2006 Jan;53(2):221-32. doi: 10.1111/j.1365-2648.2006.03718.x. PMID 16422721
- [Background] Amy NK, Aalborg A, Lyons P, Keranen L. Barriers to routine gynecological cancer screening for White and African-American obese women. Int J Obes (Lond). 2006 Jan;30(1):147-55. doi: 10.1038/sj.ijo.0803105. PMID 16231037
- [Background] Hebl MR, Xu J. Weighing the care: physicians' reactions to the size of a patient. Int J Obes Relat Metab Disord. 2001 Aug;25(8):1246-52. doi: 10.1038/sj.ijo.0801681. PMID 11477511
- [Background] Puhl RM, Brownell KD. Confronting and coping with weight stigma: an investigation of overweight and obese adults. Obesity (Silver Spring). 2006 Oct;14(10):1802-15. doi: 10.1038/oby.2006.208. PMID 17062811
- [Background] Emmer C, Bosnjak M, Mata J. The association between weight stigma and mental health: A meta-analysis. Obes Rev. 2020 Jan;21(1):e12935. doi: 10.1111/obr.12935. Epub 2019 Sep 10. PMID 31507062
- [Background] Singh K, Russell-Mayhew S, von Ranson K, McLaren L. Is there more to the equation? Weight bias and the costs of obesity. Can J Public Health. 2019 Feb;110(1):17-20. doi: 10.17269/s41997-018-0146-2. Epub 2018 Oct 26. PMID 30367387
- [Background] Hammond RA, Levine R. The economic impact of obesity in the United States. Diabetes Metab Syndr Obes. 2010 Aug 30;3:285-95. doi: 10.2147/DMSOTT.S7384. PMID 21437097
- [Background] Puhl RM, Phelan SM, Nadglowski J, Kyle TK. Overcoming Weight Bias in the Management of Patients With Diabetes and Obesity. Clin Diabetes. 2016 Jan;34(1):44-50. doi: 10.2337/diaclin.34.1.44. No abstract available. PMID 26807008
- [Background] Brown A, Flint SW, Batterham RL. Pervasiveness, impact and implications of weight stigma. EClinicalMedicine. 2022 Apr 21;47:101408. doi: 10.1016/j.eclinm.2022.101408. eCollection 2022 May. PMID 35497065
- [Background] Puhl RM, Heuer CA. Obesity stigma: important considerations for public health. Am J Public Health. 2010 Jun;100(6):1019-28. doi: 10.2105/AJPH.2009.159491. Epub 2010 Jan 14. PMID 20075322
- [Background] Puhl R, Brownell KD. Bias, discrimination, and obesity. Obes Res. 2001 Dec;9(12):788-805. doi: 10.1038/oby.2001.108. PMID 11743063
- [Background] Oliver TL, Burrell SA, Furman GE, Diewald LK, Mariani B, Starck MR, Shenkman R. Weight bias reduction intervention among nurse practitioner students using simulation-based experiences. J Am Assoc Nurse Pract. 2023 Oct 3. doi: 10.1097/JXX.0000000000000956. Online ahead of print. PMID 37788361
- [Background] Oliver TL, Qi BB, Shenkman R, Diewald L, Smeltzer SC. Weight Sensitivity Training Among Undergraduate Nursing Students. J Nurs Educ. 2020 Aug 1;59(8):453-456. doi: 10.3928/01484834-20200723-06. PMID 32757009
- [Background] Oliver TL, Qi BB, Diewald LK, Shenkman R, Kaufmann PG. Development of a weight bias reduction intervention for third-year nursing students. Clin Obes. 2022 Apr;12(2):e12498. doi: 10.1111/cob.12498. Epub 2021 Nov 25. PMID 34825503
- [Background] Batson CD, Lishner DA, Carpenter A, Dulin L, Harjusola-Webb S, Stocks EL, Gale S, Hassan O, Sampat B. "... As you would have them do unto you": Does imagining yourself in the other's place stimulate moral action? Pers Soc Psychol Bull. 2003 Sep;29(9):1190-201. doi: 10.1177/0146167203254600. PMID 15189613
- [Background] Dovidio, J.F., Gaertner, S.L., & Kawakami, K. (2003). Intergroup contact: the past, present, and future. Group Process & Intergroup Relations, 6, 25-21.
- [Background] Yoo MS, Yoo IY. The effectiveness of standardized patients as a teaching method for nursing fundamentals. J Nurs Educ. 2003 Oct;42(10):444-8. doi: 10.3928/0148-4834-20031001-06. PMID 14577730
- [Background] Johnson KV, Scott AL, Franks L. Impact of Standardized Patients on First Semester Nursing Students Self-Confidence, Satisfaction, and Communication in a Simulated Clinical Case. SAGE Open Nurs. 2020 Jun 10;6:2377960820930153. doi: 10.1177/2377960820930153. eCollection 2020 Jan-Dec. PMID 33415284
- [Background] Nagoshi MH. Role of standardized patients in medical education. Hawaii Med J. 2001 Dec;60(12):323-4. PMID 11836971
- [Background] Provider Competencies for the Prevention and Management of Obesity. (2017). Bipartisan Policy Center. Retrieved March 15, 2022, from https://bipartisanpolicy.org/library/provider-competencies-for-the-prevention-and-management-of-obesity/
- [Background] Poustchi Y, Saks NS, Piasecki AK, Hahn KA, Ferrante JM. Brief intervention effective in reducing weight bias in medical students. Fam Med. 2013 May;45(5):345-8. PMID 23681687
- [Background] O'Brien KS, Puhl RM, Latner JD, Mir AS, Hunter JA. Reducing anti-fat prejudice in preservice health students: a randomized trial. Obesity (Silver Spring). 2010 Nov;18(11):2138-44. doi: 10.1038/oby.2010.79. Epub 2010 Apr 15. PMID 20395952
- [Background] Brown, I., & Flint, S. W. (2013). Weight bias and the training of health professionals to better manage Obesity: What do we know and what should we do? Current Obesity Reports, 2(4), 333-340.
- [Background] Phelan SM, Burgess DJ, Burke SE, Przedworski JM, Dovidio JF, Hardeman R, Morris M, van Ryn M. Beliefs about the causes of obesity in a national sample of 4th year medical students. Patient Educ Couns. 2015 Nov;98(11):1446-9. doi: 10.1016/j.pec.2015.06.017. Epub 2015 Jun 27. PMID 26143579
- [Background] Foster GD, Wadden TA, Makris AP, Davidson D, Sanderson RS, Allison DB, Kessler A. Primary care physicians' attitudes about obesity and its treatment. Obes Res. 2003 Oct;11(10):1168-77. doi: 10.1038/oby.2003.161. PMID 14569041
- [Background] Alberga AS, Pickering BJ, Alix Hayden K, Ball GD, Edwards A, Jelinski S, Nutter S, Oddie S, Sharma AM, Russell-Mayhew S. Weight bias reduction in health professionals: a systematic review. Clin Obes. 2016 Jun;6(3):175-88. doi: 10.1111/cob.12147. PMID 27166133
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] Phelan SM, Burgess DJ, Yeazel MW, Hellerstedt WL, Griffin JM, van Ryn M. Impact of weight bias and stigma on quality of care and outcomes for patients with obesity. Obes Rev. 2015 Apr;16(4):319-26. doi: 10.1111/obr.12266. Epub 2015 Mar 5. PMID 25752756
- [Background] American College of Cardiology/American Heart Association Task Force on Practice Guidelines, Obesity Expert Panel, 2013. Expert Panel Report: Guidelines (2013) for the management of overweight and obesity in adults. Obesity (Silver Spring). 2014 Jul;22 Suppl 2:S41-410. doi: 10.1002/oby.20660. No abstract available. PMID 24227637
- [Background] Budd GM, Mariotti M, Graff D, Falkenstein K. Health care professionals' attitudes about obesity: an integrative review. Appl Nurs Res. 2011 Aug;24(3):127-37. doi: 10.1016/j.apnr.2009.05.001. Epub 2009 Sep 18. PMID 20974067
- [Background] World Health Organization. Weight bias and obesity stigma: considerations for the WHO European Region. (2017). Retrieved from http://www.euro.who.int/__data/assets/pdf_file/0017/351026/WeightBias.pdf?ua=1 Accessed April 23, 2022.
- [Background] Obesity Action Coalition: Understanding Obesity Stigma. (2017). Retrieved from https://4617c1smqldcqsat27z78x17-wpengine.netdna-ssl.com/wp-content/uploads/UOS_1-26-18-wo-bleed.pdf Accessed March 15, 2022.
- [Background] Puhl RM, Andreyeva T, Brownell KD. Perceptions of weight discrimination: prevalence and comparison to race and gender discrimination in America. Int J Obes (Lond). 2008 Jun;32(6):992-1000. doi: 10.1038/ijo.2008.22. Epub 2008 Mar 4. PMID 18317471
- [Background] Jastreboff AM, Kotz CM, Kahan S, Kelly AS, Heymsfield SB. Obesity as a Disease: The Obesity Society 2018 Position Statement. Obesity (Silver Spring). 2019 Jan;27(1):7-9. doi: 10.1002/oby.22378. PMID 30569641
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284